CLINICAL TRIAL: NCT02661412
Title: Immediate Loading of Implants in the Partially or Completely Edentulous Jaw
Acronym: IMLOAD
Status: Active, not recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, Maxillofacial Surgeon, Head of Department, AZ Sint-Jan AV
Other Study IDs: B049201627038
Record Dates: First submitted 2016-01-11; First posted 2016-01-22 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Jaw, Edentulous, Partially; Jaw, Edentulous
Keywords: immediate loading; biological stability; mechanical stability; long-term; marginal bone level; maxilla; immediate placement; dental implant; fibre-reinforced provisional fixed prosthesis
MeSH Terms: conditions — Jaw, Edentulous, Partially; Jaw, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to evaluate the biological and mechanical short- and long-term outcome of IL in partially or completely edentulous patients. Moreover, the investigators aim to detect potential influencing risk factors predicting undesirable prosthetic outcome.

DETAILED DESCRIPTION:
Since its introduction in the late 1990s, immediate implant loading concepts (IL) have become a frequent alternative for delayed implant procedures. IL concepts reduce chair time, the number of surgical interventions and pain, and offer instant comfort to the patient. Its reduced treatment time results in obvious socioeconomic advantages. Although there is at present abundant evidence that supports IL, evaluation of long-term biological and mechanical stability outcomes of large patient populations could allow quality improvement and more accurate patient selection. The Departments of Oral and Maxillofacial Surgery and the Department of Dentistry of the General Hospital Saint-John Bruges act as one of the pioneers of IL in Belgium, routinely performing the concept since 2001.

The investigators aim to evaluate the biological and mechanical short- and long-term outcome of IL in partially or completely edentulous patients. Moreover, the investigators aim to detect potential influencing risk factors predicting undesirable prosthetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients of all ages
* patients of all genders
* patients with partially or complete edentulous jaw
* patients treated at the department between 01/01/2001 and 31/12/2015

Exclusion Criteria:

* patients not eligible according to abovementioned criteria
* patients who required horizontal bone augmentation procedures of the complete alveolar bone
* patients who required a jaw reconstruction after tumor resection, osteoradionecrosis or medication-related osteonecrosis of the jaw

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages with loss of all or almost all teeth due to terminal periodontal disease and/or untreatable endodontic problems, that requested treatment according to the IL protocol between 01/01/2001 and 31/12/2015. Patients should have adequate bone volume to predominantly receive an implant of ≥13x3.5mm anteriorly and an implant of ≥9 x 3.5mm posteriorly. All patients, with or without a pre-prosthetic sinus floor augmentation, are included in de study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
implant survival rate | within 6 months post placement of implants
  Percentage of people in the study for which implant is still present of the fixture in the oral cavity
implant survival rate | until a maximum of 15 years of follow-up
  Percentage of people in the study for which implant is still present of the fixture in the oral cavity

SECONDARY OUTCOMES:
Infection rate | within 6 months post placement of implants
  Percentage of people in the study that develop an infection at the site of the implant in the oral cavity
Infection rate | until a maximum of 15 years of follow-up
  Percentage of people in the study that develop an infection at the site of the implant in the oral cavity
correlation between patient-mediated factors and occurrence of implant instability | within 6 months post placement of implants
  correlation between patient-mediated factors (age, gender, comorbidities, etc) and occurrence of implant instability, as clinically evaluated by the treating surgeon
correlation between patient-mediated factors and occurrence of implant instability | until a maximum of 15 years of follow-up
  correlation between patient-mediated factors (age, gender, comorbidities, etc) and occurrence of implant instability, as clinically evaluated by the treating surgeon
correlation between clinical factors and the occurrence of implant instability | within 6 months post placement of implants
  correlation between clinical factors (surgeon, surgical procedure, etc) as and the occurrence of implant instability, as clinically evaluated by the treating surgeon
correlation between clinical factors and the occurrence of implant instability | until a maximum of 15 years of follow-up
  correlation between clinical factors (surgeon, surgical procedure, etc) as and the occurrence of implant instability, as clinically evaluated by the treating surgeon
correlation between implant characteristics and occurrence of implant instability | within 6 months post placement of implants
  correlation between implant characteristics (design/finish/material) and occurrence of implant instability, as clinically evaluated by the treating surgeon
correlation between implant characteristics and occurrence of implant instability | until a maximum of 15 years of follow-up
  correlation between implant characteristics (design/finish/material) and occurrence of implant instability, as clinically evaluated by the treating surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — division of maxillofacial surgery, department of surgery, general hospital Saint-John Bruges
Locations (1):
- General Hospital Saint-John Bruges, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No